CLINICAL TRIAL: NCT01201525
Title: Pulsed Dye Laser Treatment of Recent Surgical Scars: A Prospective Single Blinded Within Patient Controlled Randomized Trial
Brief Title: Pulsed Dye Laser Treatment of Recent Surgical Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Evelien Verhaeghe, MD, University Hospital Ghent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/218
Record Dates: First submitted 2009-12-02; First posted 2010-09-14 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Surgical Scars

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical scar - part 1 (Experimental): Surgical scar - part 1
  Interventions: Procedure: Pulsed dye laser treatment
- Surgical scar - part 2 (Placebo Comparator): Surgical scar - part 2
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Pulsed dye laser treatment — Part 1 of the surgical scar will be treated with 4 595nm Pulsed dye laser treatments.
  Arms: Surgical scar - part 1
Procedure: Control — Part 2 of the surgical scar will serve as a within patient control.
  Arms: Surgical scar - part 2

SUMMARY:
Hypothesis: Improvement of recent surgical scars after treatment with 595nm Pulsed dye laser treatments.

Study design: Prospective single blinded within patient controlled randomised trial. Recent surgical scars of at least 5cm will be divided into 2 parts and randomized. 1 part will be treated with 4 595nm Pulsed dye laser treatments on a 4 weeks interval. The other part will serve as a within patient control. 1 and 6 months after the intervention both parts of the scar will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with planned surgical intervention leaving a scar from at least 5 cm in an area prone to hypertrophic scarring : neck, shoulders, chest, mandibular angle and extremities
* Age at least 18 years old.
* Patient able and willing to give written informed consent

Exclusion Criteria:

* Patients with planned surgical intervention on hands, feet and genital area
* Patients with a history of photodermatoses
* Patients with a history of keloids
* Patients with a history of adverse outcomes related to PDL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Physician global assessment for the treated and control region (PhGA) | Before start of the study, 1 and 6 months after treatment
Patient global assessment for the treated and control region (PGA) | Before start of the study, 1 and 6 months after treatment

SECONDARY OUTCOMES:
Assessment of scar color by colorimetry | Before start of the study, 1 and 6 months after treatment.
Assessment of scar tickness by ultrasound measurements | Before start of the study, 1 and 6 months after treatment.
Assessment of viscoelasticity by Cutometer measurements | Before start of the study, 1 and 6 months after treatment.
Clinical scar assessment by the Vancouver Scar scale and POSAS scale. | Before the start of the PDL treatment, and 1 and 6 months after the last treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Evelien Verhaeghe, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website of the University Hospital Ghent — http://www.uzgent.be